CLINICAL TRIAL: NCT06235424
Title: Comparison of Low Sodium Crystalloid Bretschneider-HTK Cardioplegia With Del Nido Cardioplegia in Patients Undergoing Elective Aortic Valve Replacement - a Prospective Randomized Trial
Brief Title: Del Nido Versus HTK Cardioplegia in Adult Aortic Valve Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Barbara Brzeska MD, Principal Investigator, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NKBBN/203/2018
Record Dates: First submitted 2023-12-05; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Aortic Valve Disease; Valve Disease, Heart; Cardiac Ischemia
Keywords: del Nido cardioplegia; Bretschneider HTK cardioplegia; cardioprotection; cardiac surgery; aortic valve replacement
MeSH Terms: conditions — Aortic Valve Disease; Heart Valve Diseases; Coronary Artery Disease | interventions — Del Nido cardioplegia solution; Bretschneider cardioplegic solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- del Nido cardioplegia group (Active Comparator): A group of patients that received high potassium cardioplegic solution with the addition of lidocaine, mixed with the patient's blood in 4:1 ratio
  Interventions: Drug: Del Nido Cardioplegia Solution
- Bretschneider-HTK cardioplegia group (Active Comparator): A group of patients that received low sodium cardioplegic solution with the addition of histidine, tryptophan and alpha-ketoglutarate
  Interventions: Drug: HTK solution

INTERVENTIONS:
Drug: Del Nido Cardioplegia Solution — The route of cardioplegia delivery differed according to surgeons' preferences. The total dosage of cardioplegia depends on the type of cardioplegia. The standard dose of del Nido cardioplegia in our institution is 1000 ml as an initial dose and is delivered with a system pressure of 90-150 mmHg. The solution is prepared by our hospital's pharmacy. At 60. minute of cross-clamp (XC) if XC time was expected to exceed 90 minutes another dose of solution would be delivered. The volume of an additional dose was 500 ml. The temperature of the delivered del Nido cardioplegia was 4*C.
  Other Names: del Nido; DNC
  Arms: del Nido cardioplegia group
Drug: HTK solution — The route of cardioplegia delivery differed according to surgeons' preferences. The dose of the HTK cardioplegia is calculated with an application of 20 mL/kg rule. It is delivered with a system pressure of 90-150 mmHg. If the XC time exceeds 120 minutes additional dose is given (10 mL/kg rule). The temperature of the delivered crystalloid cardioplegia is 4*C
  Other Names: HTK; Bretschneider-HTK
  Arms: Bretschneider-HTK cardioplegia group

SUMMARY:
The goal of this clinical trial is to compare del Nido and Bretschneider-HTK (HTK) cardioplegia solutions in patients undergoing elective aortic valve replacement. The main question it aims to answer is:

• Does the del Nido cardioplegia provide better cardioprotection and clinical outcomes than HTK cardioplegia? Participants will receive one of the investigated cardioplegia solutions according to the randomization.

Researchers will compare both groups in terms of cardioprotection (described as levels of CK-MB and hsTnI), in-hospital clinical outcomes, biochemical changes in coronary sinus blood and one-year follow-up.

DETAILED DESCRIPTION:
The idea of using del Nido cardioplegia in adult cardiac surgery appeared after many reports proving its safety and efficacy in the paediatric population. Therefore many adult centres started to apply it in everyday practice. Despite its growing popularity and application in different types of cardiac surgeries, there is still an insufficient number of prospective randomized trials which compare del Nido cardioplegia with the Bretschneider-HTK formula in the adult population.

The described problem will be analyzed at different levels in this prospective, randomised study.

Clinical aspects - del Nido and HTK cardioplegia will be compared in terms of intraoperative and postoperative details such as perfusion details and concentration of cardiac enzymes.

Echocardiographic changes - The next step will be revealing potential echocardiographic changes in cardiac function in short- and long-term observations after cardiac surgery.

Metabolic changes - the metabolic profile of amino acids and nucleotide changes after each cardioplegia solution delivery will be analyzed.

Statistical calculations will be performed by a qualified statistician. In the case of binary variables, Fisher's exact test will be used to assess differences between groups. In the case of quantitative variables, the compliance of the distribution with the normal distribution will be tested using the Shapiro-Wilk test. For quantitative variables with a distribution not significantly different from normal, the Student's t-test will be used for comparison between groups. If the distribution differs significantly from the normal distribution, the Mann-Whitney U test (comparisons of two samples) or the Kruskal-Wallis test (comparisons of many samples) will be used. Correlations between variables will be assessed using the Pearson or Spearman method, depending on the distribution of the variables. Repeated-measures ANOVA will be used to assess the variability of biochemical parameters over time.

In all analyses, p<0.05 will be considered as the level of statistical significance.

A comparison of the two cardioplegia solutions would allow assessing whether del Nido provides better cardioprotection than HTK.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 and over,
* qualified for elective isolated aortic valve replacement (AVR)

Exclusion Criteria:

* patients with significant coronary artery disease,
* urgent cases,
* cases with additional cardiac procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2024-09-24 (Estimated)

PRIMARY OUTCOMES:
postoperative CK-MB | measured in the 6th, 24th, and 48th hour postoperatively
  concentration of serum creatine kinase-myocardial band (CK-MB)
postoperative hsTnI | measured in the 6th, 24th, and 48th hour postoperatively
  concentration of serum high sensitive cardiac troponin I (hsTnI)

SECONDARY OUTCOMES:
CPB time | intraoperative
  Time of cardiopulmonary bypass (CPB).
XC time | intraoperative
  Time of aortic cross-clamp (XC).
Reperfusion time | intraoperative
  Time of reperfusion (between removal of cross-clamp and weaning from cardiopulmonary bypass).
Cardioplegia volume | intraoperative
  Total volume cardioplegia doses.
Cardioplegia doses | intraoperative
  Number of cardioplegia doses.
Heart rhythm after XC | intraoperative
  Type of heart rhythm after removal of aortic cross-clamp.
Need for defibrillation | intraoperative
  Need for heart defibrillations in case of ventricular fibrillation.
Number of defibrillations | intraoperative
  Number of heart defibrillations in case of ventricular fibrillation.
Intraoperative lactate concentration | intraoperative
  Lactate measured before XC, at the time of the biggest hemodilution, and after CPB.
Intraoperative pH results | intraoperative
  pH measured before XC, at the time of the biggest hemodilution, and after CPB.
Intraoperative partial pressure of oxygen | intraoperative
  Partial pressure of oxygen measured before XC, at the time of the biggest hemodilution, and after CPB.
Intraoperative partial pressure of carbon dioxide | intraoperative
  Partial pressure of carbon dioxide measured before XC, at the time of the biggest hemodilution, and after CPB.
Intraoperative base deficit | intraoperative
  Base deficit measured before XC, at the time of the biggest hemodilution, and after CPB.
Intraoperative sodium and potassium concentration | intraoperative
  Sodium and potassium concentration measured before XC, at the time of the biggest hemodilution, and after CPB.
Intraoperative amino acids concentrations | intraoperative
  Changes of amino acid concentrations in systemic and coronary sinus blood Before the procedure - sample from the peripheral arterial line before the start of the procedure.
  During cardiopulmonary bypass - samples from the peripheral arterial line and samples from the coronary sinus at 1. and 5. minute after aortic cross-clamp removal. Blood from the coronary sinus would be collected by cannula for retrograde cardioplegia delivery.
  During reperfusion - peripheral arterial line blood sample would be collected after weaning from cardiopulmonary bypass.
Intraoperative nucleotides concentrations | intraoperative
  changes of nucleotides concentrations in systemic and coronary sinus blood Before the procedure - sample from the peripheral arterial line before the start of the procedure.
  During cardiopulmonary bypass - samples from the peripheral arterial line and samples from the coronary sinus at 1. and 5. minute after aortic cross-clamp removal. Blood from the coronary sinus would be collected by cannula for retrograde cardioplegia delivery.
  During reperfusion - peripheral arterial line blood sample would be collected after weaning from cardiopulmonary bypass.
Ventilation time | 30 postoperative days
  Time of mechanical ventilation after surgery.
ICU length of stay | 30 postoperative days
  Intensive care unit (ICU) length of stay.
Hospital length of stay | 30 postoperative days
  Hospital length of stay.
Postoperative lactate concentration | 30 postoperative days
  Lactate measured at 6th, 24th, and 48th hour postoperatively.
Postoperative pH results | 30 postoperative days
  pH measured at 6th, 24th, and 48th hour postoperatively.
Postoperative partial pressure of oxygen | 30 postoperative days
  Partial pressure of oxygen measured at 6th, 24th, and 48th hour postoperatively.
Postoperative partial pressure of carbon dioxide | 30 postoperative days
  Partial pressure of carbon dioxide measured at 6th, 24th, and 48th hour postoperatively.
Postoperative base deficit | 30 postoperative days
  Base deficit measured at 6th, 24th, and 48th hour postoperatively.
Postoperative sodium and potassium levels | 30 postoperative days
  Sodium and potassium levels measured at 6th, 24th, and 48th hour postoperatively.
Maximum CRP concentration | 30 postoperative days
  Maximum C reactive protein (CRP) concentration measured during hospitalization at our institution.
Discharge CRP concentration | 30 postoperative days
  CRP results at discharge from our institution.
Maximum creatinine concentration | 30 postoperative days
  Maximum creatinine concentration measured during hospitalization at our institution.
Discharge creatinine concentration | 30 postoperative days
  Creatinine results at discharge from our institution.
Discharge Hb concentration | 30 postoperative days
  Hemoglobin (Hb) results at discharge from our institution.
Discharge Hct concentration | 30 postoperative days
  Hematocrit (Hct) results at discharge from our institution.
Discharge WBC concentration | 30 postoperative days
  White blood cells count (WBC) results at discharge from our institution.
VIS | 30 postoperative days
  Vasoactive-inotropic score (VIS) at 6th, 24th, and 48th hour postoperatively.
Rate of postoperative transfusions | 30 postoperative days
  Rate of postoperative blood product transfusions.
Rate of resternotomy | 30 postoperative days
  Rate of bleeding with the need for re-sternotomy during the early postoperative period.
Rate of pericardial drainage | 30 postoperative days
  Rate of pericardial drainages during the early postoperative period.
Rate of stroke | 30 postoperative days
  Rate of stokes during the early postoperative period.
Rate of myocardial infarction | 30 postoperative days
  Rate of myocardial infarction during the early postoperative period.
Rate of new-onset arrhythmias | 30 postoperative days
  Rate of new-onset arrhythmias (atrial fibrillation, heart block) during the early postoperative period.
In-hospital mortality rate | 30 postoperative days
  Rate of postoperative deaths that occurred during initial hospitalization.
Out-hospital mortality rate | approx one year postoperatively
  Rate of postoperative deaths that occurred after hospital discharge.
Rate of pacemaker implantation | approx one year postoperatively
  Pacemaker implantation in postoperative period.
Rate of secondary hospitalization | approx one year postoperatively
  Rate of secondary hospitalization due to late complications or other cardiac-related reasons
LVEF values changes | approx one year postoperatively
  Left ventricular ejection fraction (LVEF) will be measured during an echocardiography test before surgery, before discharge and one year after surgery.
Diastolic function changes | approx one year postoperatively
  Diastolic function measured during an echocardiography test before surgery, before discharge and one year after surgery.
2STE parameter changes | approx one year postoperatively
  2STE parameter changes (with special attention put on the ventricular septum, new hypokinetic or akinetic areas) measured during an echocardiography test before surgery, before discharge and one year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Brzeska, MD, Principal Investigator — Medical Univeristy of Gdansk
Locations (1):
- Medical University of Gdańsk, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with an interest in cardioprotection. Data or samples shared will be coded, with no PHI included.
  The data underlying this article will be shared on reasonable request.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: was not yet determined
Access Criteria: The data underlying this article will be shared on reasonable request